CLINICAL TRIAL: NCT06866938
Title: An Open Label, Single Arm Phase IIb Study of Re-treatment With [177Lu]Lu-PSMA in Men With Metastatic Castration Resistance Prostate Cancer
Brief Title: Study of Re-treatment With [177Lu]Lu-PSMA in Men With Metastatic Castration Resistance Prostate Cancer
Acronym: ReaLuP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL24_0183; 2024-512043-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic castration resistance prostate cancer; Internal vectorized radiotherapy; [177Lu]Lu-PSMA rechallenge
MeSH Terms: interventions — Pluvicto; lactitol

STUDY DESIGN:
Intervention Model Description: Prospective multicenter phase IIb single arm non randomized open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [177Lu]Lu-PSMA-617 (Experimental): Patients with metastatic castration resistance prostate cancer will be treated with intravenous [177Lu]Lu-PSMA-617 (Pluvicto, Novartis) at the dose of 7.4 GBq (±10%) every 6 weeks Treatment duration: 4 to 6 cycles (24 to 36 weeks)
  Interventions: Drug: [177Lu]Lu-PSMA-617 (Pluvicto, Novartis)

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA-617 (Pluvicto, Novartis) — Patients will be treated with intravenous [177Lu]Lu-PSMA-617 (Pluvicto, Novartis).
  One injection every 6 weeks at the dose of 7.4 GBq (±10%)

SUMMARY:
Prostate cancer is the third leading cause of cancer-related death in men in the United States and Europe. The treatment of metastatic castration-resistant prostate cancer (mCRPC) has evolved with the arrival of the radioligand [177Lu]Lu-PSMA-617, which specifically targets PSMA-expressing cancer cells.

The randomized phase III VISION study showed that [177Lu]Lu-PSMA-617 significantly improved progression-free survival and overall survival with an acceptable toxicity profile.

The ReaLuP study will evaluate the efficacy of a re-treatment of [177Lu]Lu-PSMA-617 in patients with progressive PSMA-positive mCRPC and who have been previously treated with [177Lu]Lu-PSMA without evidence of progression during this first course of treatment.

Patients will be treated until disease progression, unacceptable toxicity or death, or alternatively up to 9 months after the last dose of treatment.

At the end of this follow up period, patients will enter the " long term follow up ", at least for 2 years after the end of the last active follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 assessed within 7 days of study treatment initiation
* Histologically or cytologically confirmed adenocarcinoma of prostate (Patients with small cell carcinoma of the prostate may be included)
* Metastatic disease documented by at least one lesion on bone scan or abdominal/pelvic/chest computed tomography (CT) or magnetic resonance imaging (MRI) scan assessed by investigator. Patients without bone metastasis must have measurable lesions in extra-pelvic lymph nodes or in soft-tissues as defined by RECIST 1.1 criteria
* Confirmed progression mCRPC despite ongoing androgen deprivation with serum testosterone < 50ng/dl (1.7nM) within 3 months prior to screening. Progression is defined by the presence of at least one of the following criteria :

  * PSA progression using local laboratory values as defined by a minimum of 2 consecutive rising PSA levels with an interval of ≥1 week between each assessment where the PSA value at screening should be ≥1 ng/mL
  * Radiographic disease progression in bone based on PCWG3 criteria defined as the appearance of 2 or more new bone lesions on bone scan, with or without PSA progression
  * Radiographic disease progression in extra-pelvic lymph nodes based or soft-tissues on RECIST1.1 criteria with or without PSA progression
* PSMA positive metastatic lesions on [68Ga]-PSMA-PET/CT without PSMA negative lesion (The presence of PSMA-positive lesions is defined as [68Ga]-PSMA-11 uptake greater than that of liver parenchyma in one or more metastatic lesions of any size in any organ system. The presence of PSMA-negative lesions is defined as PSMA uptake equal to or lower than that of liver parenchyma in any lymph node with a short axis of at least 2.5 cm, in any metastatic solid-organ lesions with a short axis of at least 1.0 cm, or in any metastatic bone lesion with a soft-tissue component of at least 1.0 cm in the short axis. Patients with any PSMA negative metastatic lesion meeting these criteria are ineligible).
* Participants must have been previously treated with at least 4 consecutive cycles of [177Lu]Lu-PSMA with no evidence of progression during this first course of treatment (including radiological, clinical but also PSA progression).
* Participants must have been previously treated with at least one ARSI - Androgen Receptor Signaling Inhibitors - (including enzalutamide, apalutamide, abiraterone or darolutamide) initiated for mCSPC, nmCRPC or mCRPC. (ARSI may be also administered together with [177Lu]Lu-PSMA-617 provided that the patient has not received an identical ARSI in the past and that this ARSI was initiated at least 15 days before the first cycle of [177Lu]Lu-PSMA-617 and less than 2 months ago. The ARSI administrated in association with LuPSMA should not be considered as a prior therapy. A previous ARSI treatment is mandatory for patient eligibility)
* Patients must have been previously treated with at least one taxane based chemotherapy (with docetaxel or cabazitaxel) (The number of previously administrated lines of taxane-based therapy is not limited ; patients can have received a taxane-based chemotherapy before or after the first sequence of [177Lu]Lu-PSMA)
* Patients must have been progressed at least 120 days after the last injection of the first course of [177Lu]Lu-PSMA therapy. (Patients with a radiological or clinical progressive disease during the first 120 days after the last cycle of the first course of [177Lu]Lu-PSMA are not eligible. PSA progression is defined by a ≥ 25% increase in PSA and an absolute increase of 2 ng/mL or more from the NADIR and confirmed by a second consecutive value obtained 3 or more weeks later. Patients treated with chemotherapy, ARSI or PARP inhibitors between the first 117LuPSMA course and screening are also eligible).
* Be abstinent from heterosexual intercourse OR must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary medical cause) until 98 days (14 weeks) post-treatment.
* Adequate organ functions :

  * Bone marrow reserve :

    * ANC ≥ 1.5 X 109/L
    * Platelets ≥ 100 X 109/L
    * Hemoglobin ≥ 10 g/dL
  * Hepatic :

    * Total bilirubin ≤ 2 x ULN. For patients with known Gilbert's syndrome ≤ 3 x ULN.
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3 x ULN
  * Renal :

    * Clearance ≥40 ml/mn
* Patients must have signed informed consent prior to participating in any study related procedures
* Willing and able to comply with the protocol, including follow-up visits and examinations
* Patients have to be affiliated to the French social security system, or equivalent

Exclusion Criteria:

* History of a [177Lu]Lu-PSMA serious adverse event (SAE) or CTCAE Grade 3 or 4 AE during the initial course of [177Lu]Lu-PSMA that led to the discontinuation of treatment
* More than one course of [177Lu]Lu-PSMA therapy
* Less than 120 days from the last dose administrated in the initial course of [177Lu]Lu-PSMA treatment and the radiological or clinical disease progression, or the initiation of a subsequent therapy.
* Any history of treatment with radium-223 dichloride or other systemic radiotherapy (including strontium-89, samarium-153, actinium-PSMA...)
* Transfusion of red blood cells within 30 days prior to the first injection of the re-treatment of [177Lu]Lu-PSMA-617
* Current central nervous system (CNS) metastases
* Hypersensitivity to the active substance (Lutetium [177Lu] vipivotide tetraxetan or Gallium [68Ga] gozetotide) or to any of the excipients
* Prior > hemibody external radiotherapy
* Imminent or established spinal cord compression based on clinical findings and / or MRI that has not yet been treated
* Other malignancy treated within the last 3 years (except non-melanoma skin cancer or low-grade superficial bladder cancer)
* Chronic conditions associated with non-malignant abnormal bone growth (e.g., confirmed Paget's disease of bone)
* Ongoing participation in any other clinical trial who may interfere with the present study in the judgment of the investigator
* Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.
* Active clinically significant cardiac disease
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study
* Patients under tutorship or guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival rate | At 24 weeks after the start of study treatment
  Proportion (in %) of patients alive without disease progression at 24 weeks. Progression is defined by imaging (bone scan and CT-scan) according to RECIST 1.1 and/or PCWG3 criteria.

SECONDARY OUTCOMES:
Imaging-based radiographic progression (rPFS) | Through study completion, a maximum of 57 months
  Imaging-based radiographic progression defined as the time from the first cycle of re-treatment to the date of radiographic disease progression or death from any cause.
Overall survival | Through study completion, a maximum of 57 months
  Overall Survival (Os) defined as the time from the first cycle of re-treatment to the date of death from any cause
Objective response rate | Through study completion, a maximum of 57 months
  Objective response rate (ORR) (Complete Response (CR) + Partial Response (PR)) measured by RECIST v1.1 response.
Duration of response | Through study completion, a maximum of 57 months
  Duration of response (DOR) will be measured in patients who achieved a CR or PR between the date of first response and the date of RECIST progression or death.
Disease Control Rate | Through study completion, a maximum of 57 months
  Disease control rate as measured by RECIST v1.1 response. Rates will be measured in soft tissue, lymph nodes and visceral lesions.
Progression free survival | Through study completion, a maximum of 57 months
  Progression free survival will be defined as the date of first cycle of [177Lu]Lu-PSMA-617 re-treatment to the date of first evidence of radiographic progression, clinical progression, PSA progression, or death from any cause, whichever occurs first.
Biological response | Through study completion, a maximum of 57 months
  Proportion of participants with a PSA response defined as a patient who has achieved a ≥ 50% PSA decrease from baseline that is confirmed with a second PSA measurement at ≥ 4 weeks.
Time to PSA progression | Through study completion, a maximum of 57 months
  Time to PSA progression will be defined as the date from first cycle of [177Lu]Lu-PSMA-617 re-treatment to a ≥ 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir and confirmed by a second consecutive value obtained 3 or more weeks later. Where no decline from baseline is documented, PSA progression is defined as a 25% increase from the baseline value along with an increase in absolute value of 2 ng/mL or more after 12 weeks of treatment.
Safety : Adverse Events | Through study completion, a maximum of 57 months
  Safety of re-treatment will be assessed by percentage of patients with all grade and Serious AEs; percentage of patients with SAEs during the active follow up period; percentage of patients with an interruption of [177Lu]Lu-PSMA-617 re-treatment; Percentage of patients who discontinue [177Lu]Lu-PSMA-617 re-treatment secondary to an AEs or death; Number and grade of AE related to the investigational medicinal product or to the procedures added by the research
Pain assessment | Up to 6 weeks from the last [177Lu]Lu-PSMA-617 administration
  Pain will be assessed with the BPI-SF (Brief Pain Inventory - Short Form) questionnaire.
  BPI-SF is a multidimensional scale evaluating the intensity and the interference of pain in life activities: four pain severity items and seven pain interference items rated on 0-10 scales, and the question about percentage of pain relief by analgesics.
  Pain severity: The BPI assesses pain at its "worst," "least," "average," and "now" (current pain); each of the forth items are used singly to represent pain severity.
  Pain interference: The BPI measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is typically scored as the mean of the seven interference items. This mean can be used if more than 50%, or four of seven, of the total items have been completed on a given administration.
  The highest is the score, the worst are the pain and pain interference
Quality of life assessment | Up to 6 weeks from the last [177Lu]Lu-PSMA-617 administration
  Aspects of HRQoL will be reported using Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire.
  FACT-P score range 0-156; the higher the score, the better the QoL Subscales: Physical well-being (0-28) Social/Family well-being (0-28) Emotional well-being (0-24) Functional well-being (0-28) Prostate cancer subscale (0-48)
Symptomatic Skeletal Event (SSE) assessment | Through study completion, a maximum of 57 months
  Time to first symptomatic skeletal event (SSE) and SSE-free survival defined as date of first injection of [177Lu]Lu-PSMA-617 re-treatment to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, or requirement for radiation therapy to relieve bone pain, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Médecine Nucléaire, Institut Bergonié, Bordeaux
  - Oncologie Médicale, CHU Brest-Hôpital Morvan, Brest
  - Hôpital Louis Pradel, Hospices Civils de Lyon, Bron
  - Oncologie Médicale, Centre François Baclesse, Caen
  - Oncologie Médicale, Centre Jean Perrin, Clermont-Ferrand
  - Médecine Nucléaire, Centre Hospitalier de Grenoble Alpes, Grenoble
  - Médecine Nucléaire, Centre Léon Berard, Lyon
  - Médecine Nucléaire, CHU de Nantes Hôtel-Dieu, Nantes
  - Oncologie Médicale, Centre Antoine Lacassagne, Nice
  - Institut de cancérologie du Gard, Nîmes
  - Oncologie Médicale, Centre Hospitalier Lyon Sud, HCL, Pierre-Bénite
  - Oncologie Médicale, Centre Henri Becqueret, Rouen
  - Oncologie Médicale, CHU Saint Etienne, Saint-Priest-en-Jarez
  - Médecine Nucléaire, Institut de Cancérologie de Strasbourg, Strasbourg
  - CHU de Nancy, Vandœuvre-lès-Nancy
  - Médecine Nucléaire, Institut Gustave Roussy, Villejuif